CLINICAL TRIAL: NCT04574531
Title: Comparative Study of US Elastography and Color Doppler US in Differentiating Breast Masses in Correlation to Histopathology
Brief Title: us Elastography and us Doppler in Differentiating Breast Masses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Sayed Mohamed Abd Elsamie, Comparative study of US elastography and color Doppler US in differentiating breast masses in correlation to histopathology, Assiut University
Other Study IDs: breast US elastography
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Breast Lump (Malignant)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to compare the diagnostic performance of grey scale US , US elastography & color Doppler US in differentiating breast masses comparable with histopathology as a gold standard.

DETAILED DESCRIPTION:
Breast cancer is the most fre¬quently diagnosed cancer and the chief cause of cancer death among women worldwide, with an es¬timated 1.7 million cases.

Breast cancer alone accounts for 25% of all cancer cases and 15% of all cancer deaths among females .so, Its high incidence has led to research on new diagnostic imaging techniques for early diagnosis and to improve patient's mortality rate[1].

Application of imaging techniques together with other investigation would help clinical decision making. the most important factor in reducing mortality of certain cancers is an early diagnosis of cancer via screening based on imaging[2].

US is an accurate method for detection of breast masses ; however, US has a low accuracy in differentiating between benign from malignant breast masses . US could suggest a malignancy likelihood criteria of a breast mass, such as hypoechogenicity, irregular margins, microcalcifications, increased vascularity by Doppler and us elastography [3].

Ultrasound elastography provides a non-invasive evaluation of the "stiffness" of a lesion. Recent studies show that ultrasonographic elastogra¬phy (USE) provides higher diagnostic accuracy together with Doppler application compared with conventional B-mode ultrasonography during breast cancer diagnosis, which eventually helps to reduce false-positive results (ie, increased specificity) and therefore is useful in avoiding breast biopsy[4].

US elastography has been used to detect the nature of breast lesions , by measuring the tissue stiffness non invasively. It depends on tissue deformation strain that is caused by external compression. it is complementary to gray scale findings particularly in lesions with indeterminate US findings, also US elastography could be used to guide the follow up of leisons diagnosed as benign at ( FNA) fine needle aspiration.[5][6]

ELIGIBILITY:
Inclusion Criteria:

* patients with breast masses referred to our department of diagnostic radiology for radiological assessment.

Exclusion Criteria:

Patients with purely cystic lesions on conventional breast ultrasound. Breast implant. Superficial lesions (>5 mm deep to skin surface).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will subjected to :
  Full history taking, clinical examination by referring physician . Then the patient will be examined by Gray scale US , doppler and elastography at Radiology department.
  On Gray scale:Echogenicity of the mass with respect to normal breast parenchyma, diameter A/T ,margins and calcifications.
  While on Color Doppler, to describe the vascular patterns. Masses and axillary lymph nodes (if detected) will be identified as nonvascular or vascular (peripheral, central, or mix).
  (A) Strain elastography Color coding is classified into 5 groups according to the Ueno classification, score one (softest component) and score five (hardest component) .
  (B) Shear wave elastography A ROI rectangular box was adjusted on the observed target lesion including sufficient amount of surrounding healthy breast tissue.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
comparison between us elastography and doppler us of breast masses with the histopathology of the specimens | baseline
  comparitive study between us elastography and doppler us of breast masses in differentiating breast masses

REFERENCES:
- [Background] Sigrist RMS, Liau J, Kaffas AE, Chammas MC, Willmann JK. Ultrasound Elastography: Review of Techniques and Clinical Applications. Theranostics. 2017 Mar 7;7(5):1303-1329. doi: 10.7150/thno.18650. eCollection 2017. PMID 28435467
- [Background] Barr RG. Breast Elastography: How to Perform and Integrate Into a "Best-Practice" Patient Treatment Algorithm. J Ultrasound Med. 2020 Jan;39(1):7-17. doi: 10.1002/jum.15137. Epub 2019 Oct 16. PMID 31617225